CLINICAL TRIAL: NCT05432323
Title: Multi-family Therapy and School Refusal: an Exploratory Study With Adolescents and Their Families
Acronym: Multi-Fast
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211594; 2021-A01853-38 (Other: France : national drug safety agency)
Record Dates: First submitted 2022-06-14; First posted 2022-06-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: School Phobia
Keywords: Adolescence; School Phobia; Multi-family therapy; Anxiety disorder
MeSH Terms: conditions — Phobia, School; Anxiety Disorders | interventions — Psychotherapy, Group

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adolescents
  Interventions: Behavioral: Multi-family therapy
- Parents
  Interventions: Behavioral: Multi-family therapy

INTERVENTIONS:
Behavioral: Multi-family therapy — 8 sessions of Multi-family therapy of 3 hours each during 24 weeks

SUMMARY:
The purpose of this study is to determine whether multi-family therapy is effective in the treatment of school refusal with anxiety in adolescence.

DETAILED DESCRIPTION:
Anxious school refusal in adolescence is a major public health problem. The involvement of families is essential and multi-family therapy has shown its effectiveness for many mental disorders. This study aims to explore the benefit of multi-family therapy in the care of anxious school refusal in adolescence.

The method will be qualitative with phenomenological analysis of semi-structured interviews with adolescents and their parents and quantitative with a SCED design to assess the evolution of the level of anxiety of adolescents and parents, as well as personalized objectives.

The objective is therefore to improve the care of adolescents with anxious school refusal.

ELIGIBILITY:
Inclusion Criteria:

* Families with an adolescent
* Aged 12 to 18
* Totally out of school for more than 2 consecutive weeks and less than 18 months
* Follow-up at the Maison de Solenn-Maison des Adolescents (Cochin Hospital AP-HP) for a school refusal
* Having agreed to participate in a multi-family therapy
* Domiciliation in Ile de France
* Agreement of the parents and the adolescent to participate in the study: Collection of the non-opposition of non-emancipated minors and their legal representatives

Exclusion Criteria:

* any family situation that makes it impossible to bring parents and children together in family therapy
* patient under curatorship or tutorship
* patient with AME (french State Medical Aid)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cochin Hospital, Maison de Solenn-Maison des Adolescents, Paris, AP-HP Primary care clinic, Day care clinic
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 13 to 15 months
  Visual Analogue Scale for anxiety (adolescents and parents) / 0 = no anxiety at all, 10 = maximum anxiety imaginable / Weekly measurement between inclusion and the end of the Single Case Experimental Design (SCED) follow-up (13 to 15 months)

SECONDARY OUTCOMES:
Goal Attainment Scale (GAS) | 13 to 15 months
  School attendance (adolescent) / 3-terminal GAS are 5-level GAS, i.e. with a possible rating ranging from -2 to +2. Level -2 corresponds to the initial state at the time of inclusion. Levels -2, 0 and +2 are precisely described, level -1 corresponds to a rating between -2 and 0 and level +1 to a rating between 0 and +2 / Weekly measurements, parents and adolescent, once a week from inclusion to the end of the SCED follow-up (13 to 15 months)
Adolescent Depression Rating Scale (ADRS) | 13 to 15 months
  Depression (adolescent) / 10 questions / Monthly measurements, adolescent and referring psychiatrist once a month from inclusion to the end of the SCED follow-up (13 to 15 months)
Family Assessment Device General Functioning (FAD-GF) | 13 to 15 months
  Family functioning / 12 questions, minimum = 12, maximum = 48 / Monthly measurements, parents and adolescent, once a month from inclusion to the end of the SCED follow-up (13 to 15 months)
Global Assessment of Functioning Scale (GAF) | 13 to 15 months
  Global Functioning of the adolescent / From 0 = inadequate information, to 100 = higher level of functioning in a wide variety of activities - V-axis of the DSM 5 / Monthly measurements, referring psychiatrist, once a month from inclusion to the end of the SCED follow-up (13 to15 months)
CSQ 8 (Client Satisfaction Questionnaire) | 7 to 9 months
  Satisfaction of the patients and the parents with multi-family therapy / 8 questions, minimum score = 8, maximum = 32 / At the end of the multifamily therapy, parents and teenager
Semi-structured interview | 7 to 9 months
  Semi-structured interview with qualitative phenomenological analysis (patients and parents) At the end of multi-family therapy
Semi-structured interview | 19 to 21 months
  Semi-structured interview with qualitative phenomenological analysis (patients and parents) 12 months after the end of multi-family therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Rose MORO, MD, PhD, PU-PH, Study Director — Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP); Aurélie HARF, MD, PhD, Principal Investigator — Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP)
Locations (1):
- Maison de Solenn Maison des Adolescents, Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No